CLINICAL TRIAL: NCT00694109
Title: An Open-label Extension Study to Assess the Long-term Safety and Efficacy of ISIS 301012 in Patients With Familial Hypercholesterolemia or Severe-Hypercholesterolemia
Brief Title: An Open-label Extension Study to Assess the Long-term Safety and Efficacy of ISIS 301012 (Mipomersen) in Patients With Familial Hypercholesterolemia or Severe-Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 301012-CS6; 2005-003450-10 (EudraCT Number)
Record Dates: First submitted 2008-06-05; First posted 2008-06-10 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-08

CONDITIONS: Lipid Metabolism, Inborn Errors; Hypercholesterolemia, Autosomal Dominant; Hyperlipidemias; Metabolic Diseases; Hyperlipoproteinemia Type II; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Metabolic Disorder; Congenital Abnormalities; Hypercholesterolemia; Hyperlipoproteinemias; Dyslipidemias; Lipid Metabolism Disorders
Keywords: Familial Hypercholesterolemia; FH; Heterozygous Familial Hypercholesterolemia; HeFH; Homozygous Familial Hypercholesterolemia; HoFH
MeSH Terms: conditions — Lipid Metabolism, Inborn Errors; Hyperlipoproteinemia Type II; Hyperlipidemias; Metabolic Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Congenital Abnormalities; Hypercholesterolemia; Hyperlipoproteinemias; Dyslipidemias; Lipid Metabolism Disorders; Homozygous Familial Hypercholesterolemia | interventions — mipomersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mipomersen (Experimental): Mipomersen Sodium once a week for up to 4 years (depending on participant's consent). Participants were followed for additional 24 week post-treatment.
  Interventions: Drug: Mipomersen Sodium

INTERVENTIONS:
Drug: Mipomersen Sodium — Subcutaneous injection as a single injection directly into the abdomen, thigh, or outer area of the upper arm.
  Other Names: ISIS 301012; Kynamro®

SUMMARY:
To evaluate the safety and efficacy of extended dosing with mipomersen (ISIS 301012) in participants with familial hypercholesterolemia or severe hypercholesterolemia on lipid-lowering therapy who had completed either the 301012-CS5 (NCT00607373), 301012-CS7 (NCT00706849), 301012-CS17 (NCT00477594) or MIPO3500108 (NCT00794664) clinical drug trials.

DETAILED DESCRIPTION:
All familial hypercholesterolemia (FH) or severe hypercholesterolemia participants who had tolerated the treatment regimen in Protocol 301012-CS5 (NCT00607373), 301012-CS7 (NCT00706849) or MIPO3500108 (NCT00794664) and satisfactorily completed the study through to Week 28 were eligible for participation in this open label treatment extension study for up to 4 years or until mipomersen was commercially available, whichever comes first. Consenting participants who had tolerated mipomersen and satisfactorily completed 301012-CS17 (NCT00477594) through Year 3 may also enroll for up to an additional 2 years of treatment in this study or until mipomersen was commercially available, whichever comes first. All participants, who entered the study, received 200 mg mipomersen (ISIS 301012) subcutaneously (s.c.) every week, including those who were randomized to placebo in their initial study. Participants who were originally enrolled in Protocol 301012-CS5 (NCT00607373) and weighed <50 kg received 160 mg every week. Dose adjustments (70 mg injections administered three times per week, on separate days) were allowed for participants who were not tolerating or who had previous issues with tolerating the once a week injections due to injection site reactions (ISRs) or flu-like symptoms. Study visits and clinical lab assessments including hematology with differential, chemistry, serum lipid panel (total cholesterol, LDL-C, very low density lipoprotein cholesterol (VLDL-C), high density lipoprotein cholesterol (HDL-C), apolipoprotein B (apoB), apoA-1, triglycerides (TG) and Lp(a), and urinalysis was to be performed every 4-10 weeks during the treatment period. Plasma trough mipomersen (ISIS 301012) levels was to be measured to estimate exposure. Participants who completed dosing or who discontinued prematurely from the study for any reason was followed for safety for 24 weeks (safety follow-up period) after their last dose of mipomersen (ISIS 301012) or longer in the case of a significant adverse events (AE) or abnormal biochemical or clinical finding. Participants were required to return to the study center for clinical evaluation and clinical laboratory tests every 8 weeks during the safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Satisfactory completion of dosing in their initial study (Protocol 301012-CS5 [NCT00607373], 301012-CS7 [NCT00706849], 301012-CS17 [NCT00477594], or MIPO3500108 [NCT00794664])

Exclusion Criteria:

* Had any new condition or worsening of existing condition which in the opinion of the Investigator would make the participant unsuitable for enrollment, or could interfere with the participant participating in or completing the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2008-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (32):
- United States (20):
  - Mission Viejo, California
  - Newport Beach, California
  - Bridgeport, Connecticut
  - Melbourne, Florida
  - Winter Park, Florida
  - Chicago, Illinois
  - Kansas City, Kansas
  - Biddeford, Maine
  - Boston, Massachusetts
  - St Louis, Missouri
  - Concord, New Hampshire
  - New York, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Franklin, Ohio
  - Portland, Oregon
  - Nashville, Tennessee
  - Dallas, Texas
  - Seattle, Washington
- São Paulo, São Paulo, Brazil
- Canada (6):
  - Winnipeg, Manitoba
  - London, Ontario
  - Chicoutimi, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
- Singapore, Singapore
- South Africa (2):
  - Observatory, South Africa
  - Parktown, South Africa
- Taipei, Taiwan, Taiwan
- London, United Kingdom, United Kingdom

REFERENCES:
- [Derived] Duell PB, Santos RD, Kirwan BA, Witztum JL, Tsimikas S, Kastelein JJP. Long-term mipomersen treatment is associated with a reduction in cardiovascular events in patients with familial hypercholesterolemia. J Clin Lipidol. 2016 Jul-Aug;10(4):1011-1021. doi: 10.1016/j.jacl.2016.04.013. Epub 2016 May 9. PMID 27578134
- [Derived] Santos RD, Duell PB, East C, Guyton JR, Moriarty PM, Chin W, Mittleman RS. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J. 2015 Mar 1;36(9):566-75. doi: 10.1093/eurheartj/eht549. Epub 2013 Dec 23. PMID 24366918

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 33 centers in 7 countries. A total of 144 patients were enrolled in the study. 1 patient never received study drug. 2 of the enrolled patients came from a phase 2 study and its extension and consequently had very different treatment from the other treated patients, and thus were excluded from all summary tables.
Pre-assignment Details: Participants who successfully completed ISIS 301012 CS5 (NCT00607373), ISIS 301012CS7 (NCT00706849), ISIS 301012CS17 (NCT00694109) or MIPO3500108 (NCT00794664) with an acceptable safety profile were eligible for study.
Groups:
- Mipomersen: Mipomersen Sodium 200 mg (for participants weighed ≥ 50 kg) or 160 mg (for participants weighed <50 kg) subcutaneous injection once a week for up to 4 years (depending on participant's consent). Participants were followed for additional 24 week post-treatment.
Period: Overall Study
Arm/Group | Mipomersen
Started | 142 (This does not include 2 patients from phase 2 trial with very different treatment experience.)
Treated | 141
Consented 2 Years Additional Treatment | 42
Completed Consented Length of Treatment | 60
Completed | 25
Not Completed | 117
Not completed — Physician Decision | 3
Not completed — Adverse Event | 74
Not completed — Not consent of more 2 years of treatment | 18
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 13
Not completed — Pregnancy | 1
Not completed — Enrolled but not treated | 1
Not completed — Other | 2
Not completed — Consented but no additional treatment | 3

BASELINE CHARACTERISTICS:
Population: Safety set: All enrolled participants who received at least 1 injection of study drug.
Arm/Group | Mipomersen
Number analyzed (Participants) | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 84

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C)
Description: Baseline was defined as the last value prior to receiving the first dose of mipomersen in this study (for participants randomized to placebo in their index study and for participants randomized to mipomersen in their index study and their first dose of mipomersen in this study was administered >=6 months from their last dose of mipomersen in their index study), or the last value prior to receiving the first dose of mipomersen in their index study (for participants randomized to mipomersen in their index study and their first dose of mipomersen in this study was administered <6 months from their last dose of mipomersen in their index study).
Time Frame: Baseline up to Week 234; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 141
percent change
  week 26 (n = 130) | -28.5 [-31.9 to -25.1]
  week 52 (n = 111) | -27 [-31.2 to -22.8]
  week 76 (n = 66) | -27.3 [-33 to -21.6]
  week 104 (n = 57) | -27.9 [-33.9 to -21.8]
  week 130 (n = 42) | -21.9 [-31.1 to -12.7]
  week 156 (n = 30) | -21.4 [-31.2 to -11.7]
  week 182 (n = 26) | -23.6 [-36.6 to -10.6]
  week 208 (n = 27) | -26.3 [-36.4 to -16.2]
  week 234 (n = 17) | -22.5 [-34.3 to -10.6]
  24 weeks post last dose (n=117) | 1.6 [-2.6 to 5.9]

2. Primary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B)
Description: as for outcome 1
Time Frame: Baseline up to Week 234; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 141
percent change
  week 26 (n = 130) | -28.9 [-32 to -25.8]
  week 52 (n = 111) | -28.1 [-32 to -24.2]
  week 76 (n = 66) | -30.3 [-34.7 to -26]
  week 104 (n = 57) | -31.2 [-36.5 to -25.9]
  week 130 (n = 43) | -29.1 [-35.7 to -22.5]
  week 156 (n = 30) | -30.2 [-38.1 to -22.2]
  week 182 (n = 26) | -31.1 [-39.9 to -22.2]
  week 208 (n = 27) | -33.3 [-40.8 to -25.9]
  week 234 (n = 17) | -31.4 [-38.7 to -24.1]
  24 weeks post last dose (n=117) | -3.46 [-6.9 to 0]

3. Primary Outcome: Percent Change From Baseline in Total Cholesterol
Description: as for outcome 1
Time Frame: Baseline up to Week 234; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 141
percent change
  week 26 (n = 130) | -21.7 [-24.4 to -18.9]
  week 52 (n = 111) | -20.4 [-23.9 to -16.8]
  week 76 (n = 66) | -20.1 [-24.6 to -15.5]
  week 104 (n = 57) | -19.8 [-24.8 to -14.7]
  week 130 (n = 43) | -14.9 [-22.1 to -7.8]
  week 156 (n = 30) | -14.4 [-22.3 to -6.6]
  week 182 (n = 26) | -14.3 [-25 to -3.5]
  week 208 (n = 27) | -16.5 [-24.2 to -8.8]
  week 234 (n = 17) | -12.5 [-21.5 to -3.4]
  24 weeks post last dose (n=117) | 1.94 [-1.5 to 5.4]

4. Primary Outcome: Percent Change From Baseline in Non High Density Lipoprotein Cholesterol (Non-HDL-C)
Description: as for outcome 1
Time Frame: Baseline up to Week 234; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 141
percent change
  week 26 (n = 130) | -27.2 [-30.4 to -24.1]
  week 52 (n = 111) | -25.4 [-29.5 to -21.3]
  week 76 (n = 66) | -25 [-30.4 to -19.7]
  week 104 (n = 57) | -26.2 [-32 to -20.4]
  week 130 (n = 43) | -20.7 [-29.1 to -12.3]
  week 156 (n = 30) | -20 [-29.6 to -10.3]
  week 182 (n = 26) | -21.7 [-34.7 to -8.7]
  week 208 (n = 27) | -23.9 [-33.7 to -14.1]
  week 234 (n = 17) | -19.9 [-31.5 to -8.2]
  24 weeks post last dose (n=117) | 2.5 [-1.8 to 6.7]

5. Secondary Outcome: Percent Change From Baseline in Triglycerides
Description: as for outcome 1
Time Frame: Baseline up to Week 234; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 141
percent change
  week 26 (n = 130) | -20.1 [-33.1 to -1.2]
  week 52 (n = 111) | -7.9 [-31.5 to 16.9]
  week 76 (n = 66) | -10.2 [-27.7 to 13.8]
  week 104 (n = 57) | -12.5 [-37.1 to 7.2]
  week 130 (n = 43) | -10.9 [-36 to 10]
  week 156 (n = 30) | -10.4 [-23.8 to 12.7]
  week 182 (n = 26) | -12.9 [-27.4 to -1.6]
  week 208 (n = 27) | -13.9 [-40 to 33]
  week 234 (n = 17) | 1.3 [-15.4 to 15.7]
  24 weeks post last dose (n=117) | 2.1 [-17.2 to 27.7]

6. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a)
Description: as for outcome 1
Time Frame: Baseline up to Week 234; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 141
percent change
  week 26 (n = 130) | -20.5 [-39.3 to -3.6]
  week 52 (n = 111) | -19 [-33.3 to 0]
  week 76 (n = 66) | -17.9 [-33.3 to -0.5]
  week 104 (n = 57) | -16.6 [-36.1 to 0]
  week 130 (n = 43) | -15.8 [-31.3 to 0]
  week 156 (n = 30) | -9.1 [-33.8 to 7.3]
  week 182 (n = 26) | -9 [-27.2 to 7.6]
  week 208 (n = 27) | -9.9 [-32.5 to 4.1]
  week 234 (n = 17) | -18.3 [-31.6 to -4.8]
  24 weeks post last dose (n=117) | 0 [-6 to 5]

7. Secondary Outcome: Percent Change From Baseline in LDL Particles' Size (Total)
Description: as for outcome 1
Time Frame: Baseline up to End of treatment; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time. Number of participants analyzed = participants with available data for LDL Particles' Size (Total).
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 140
percent change
  week 52 (n = 91) | -26.77 [-32.7 to -20.8]
  week 104 (n = 47) | -27.77 [-35.3 to -20.3]
  week 156 (n = 20) | -25.1 [-40.3 to -9.9]
  week 208 (n = 19) | -32.65 [-44.9 to -20.4]
  End of treatment (n=139) | -22.63 [-27 to -18.3]
  24 weeks post last dose (n=115) | 6.11 [0.8 to 11.5]

8. Secondary Outcome: Percent Change From Baseline in LDL Particles' Size (Large)
Description: as for outcome 1
Time Frame: Baseline up to End of treatment; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time. Number of participants analyzed = participants with available data for LDL Particles' Size (Large).
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 140
percent change
  week 52 (n = 91) | -5.01 [-16.8 to 6.8]
  week 104 (n = 47) | -14.32 [-27 to -1.6]
  week 156 (n = 20) | -27.04 [-40.6 to -13.4]
  week 208 (n = 19) | -22.67 [-41.6 to -3.8]
  End of treatment (n=139) | -2.94 [-13.2 to 7.3]
  24 weeks post last dose (n=115) | 6.19 [-6.1 to 18.5]

9. Secondary Outcome: Percent Change From Baseline in LDL Particles' Size (Medium)
Description: as for outcome 1
Time Frame: Baseline up to End of treatment; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time. Number of participants analyzed = participants with available data for LDL Particles' Size (Medium).
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 140
percent change
  week 52 (n = 91) | -9.50 [-31.8 to 12.8]
  week 104 (n = 47) | 11.09 [-42.2 to 64.4]
  week 156 (n = 20) | -19.62 [-57.3 to 18]
  week 208 (n = 19) | -15.82 [-62 to 30.4]
  End of treatment (n=139) | -5.65 [-30.3 to 19]
  24 weeks post last dose (n=115) | 46.92 [5.6 to 88.2]

10. Secondary Outcome: Percent Change From Baseline in LDL Particles' Size (Small)
Description: as for outcome 1
Time Frame: Baseline up to End of treatment; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time. Number of participants analyzed = participants with available data for LDL Particles' Size (Small).
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 140
percent change
  week 52 (n = 91) | -8.79 [-33.7 to 16.2]
  week 104 (n = 47) | 1.72 [-43.9 to 47.4]
  week 156 (n = 20) | -18.95 [-58.8 to 20.9]
  week 208 (n = 19) | -27.95 [-67.9 to 12]
  End of treatment (n=139) | -5.17 [-29.2 to 18.8]
  24 weeks post last dose (n=115) | 51.94 [7.7 to 96.2]

11. Secondary Outcome: Percent Change From Baseline in LDL Particles' Size (Very Small)
Description: as for outcome 1
Time Frame: Baseline up to End of treatment; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time. Number of participants analyzed = participants with available data for LDL Particles' Size (Very Small).
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 140
percent change
  week 52 (n = 91) | -5.05 [-32.2 to 22.2]
  week 104 (n = 47) | -0.11 [-44.4 to 44.2]
  week 156 (n = 20) | -18.7 [-59.2 to 21.8]
  week 208 (n = 19) | -30.77 [-69.3 to 7.8]
  End of treatment (n=139) | 0.75 [-28 to 29.5]
  24 weeks post last dose (n=115) | 60.22 [7.5 to 112.9]

12. Secondary Outcome: Percent Change From Baseline in HDL Particles' Size (Large)
Description: as for outcome 1
Time Frame: Baseline up to End of treatment; 24 weeks post treatment (up to 4.5 years)
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 140
percent change
  week 52 (n = 89) | 160.8 [-38.3 to 359.9]
  week 104 (n = 47) | 43.23 [-12.2 to 98.7]
  week 156 (n = 20) | 58.26 [-38 to 154.6]
  week 208 (n = 19) | 61.76 [-41.6 to 165.2]
  End of treatment (n=134) | 121.16 [-17.3 to 259.6]
  24 weeks post last dose (n=110) | 85.93 [-7.3 to 179.1]

13. Secondary Outcome: Percent Change From Baseline in HDL Particles' Size (Medium)
Description: as for outcome 1
Time Frame: Baseline up to End of treatment; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time. Number of participants analyzed = participants with available data for HDL Particles' Size (Medium).
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 140
percent change
  week 52 (n = 44) | 154.77 [2.8 to 306.8]
  week 104 (n = 28) | 176.14 [-68.6 to 420.9]
  week 156 (n = 9) | 21.24 [-65.1 to 107.6]
  week 208 (n = 8) | 838.32 [-1109.3 to 2785.9]
  End of treatment (n= 68) | 388.16 [94.5 to 681.8]
  24 weeks post last dose (n=56) | 233.78 [7.9 to 459.7]

14. Secondary Outcome: Percent Change From Baseline in HDL Particles' Size (Small)
Description: as for outcome 1
Time Frame: Baseline up to End of treatment; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time. Number of participants analyzed = participants with available data for HDL Particles' Size (Small).
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 140
percent change
  week 52 (n = 91) | 1.83 [-7.3 to 10.9]
  week 104 (n = 47) | -9.81 [-17.7 to -2]
  week 156 (n = 20) | -14.18 [-25.1 to -3.2]
  week 208 (n = 19) | -11.47 [-20 to -2.9]
  End of treatment (n= 139) | 0.44 [-6.9 to 7.7]
  24 weeks post last dose (n=115) | 8.31 [0.6 to 16]

15. Secondary Outcome: Percent Change From Baseline in Intermediate Density Lipoprotein Particles' Size
Description: as for outcome 1
Time Frame: Baseline up to End of treatment; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time. Number of participants analyzed = participants with available data for Intermediate Density Lipoprotein Particles' Size.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 140
percent change
  week 52 (n = 79) | -9.9 [-45.6 to 25.8]
  week 104 (n = 40) | -27.35 [-66.5 to 11.8]
  week 156 (n = 16) | 155.42 [-90.1 to 401]
  week 208 (n = 15) | 32.88 [-104 to 169.8]
  End of treatment (n= 122) | 24.66 [-28.4 to 77.8]
  24 weeks post last dose (n=101) | 57.46 [15.2 to 99.8]

16. Secondary Outcome: Percent Change From Baseline in Very Low Density Lipoprotein (VLDL) Particles' Size (Large) and Chylomicron Particles' Size
Description: as for outcome 1
Time Frame: Baseline up to End of treatment; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time. Number of participants analyzed = participants with available data for Very Low Density Lipoprotein (VLDL) Particles' Size (Large) and Chylomicron Particles' Size.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 140
percent change
  week 52 (n = 86) | 109.23 [33.7 to 184.8]
  week 104 (n = 46) | 107.5 [-10.2 to 225.2]
  week 156 (n = 19) | 123.42 [-113 to 359.8]
  week 208 (n = 18) | 241.76 [-241.5 to 725.1]
  End of treatment (n= 132) | 86.75 [28.4 to 145.1]
  24 weeks post last dose (n=110) | 90.82 [21.8 to 159.9]

17. Secondary Outcome: Percent Change From Baseline in VLDL Particles' Size (Medium)
Description: as for outcome 1
Time Frame: Baseline up to End of treatment; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time. Number of participants analyzed = participants with available data for VLDL Particles' Size (Medium).
Measure: Mean (95% Confidence Interval); unit: percent change
Groups:
- Mipomersen: Mipomersen Sodium 200 mg (for participants weighed ≥ 50 kg) or 160 mg (for participants weighed <50 kg) once a week subcutaneously for up to 4 years (depending on participant's consent). Participants were followed for additional 24 week post-treatment.
Arm/Group | Mipomersen
Number analyzed (Participants) | 140
percent change
  week 52 (n = 88) | 70.81 [2.1 to 139.5]
  week 104 (n = 47) | 97.74 [-21 to 216.5]
  week 156 (n = 20) | 172.46 [5.3 to 339.7]
  week 208 (n = 19) | 98.7 [-71.3 to 268.7]
  End of treatment (n= 136) | 63.25 [12.1 to 114.4]
  24 weeks post last dose (n=113) | 99.57 [16.8 to 182.3]

18. Secondary Outcome: Percent Change From Baseline in VLDL Particles' Size (Small)
Description: as for outcome 1
Time Frame: Baseline up to End of treatment; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time. Number of participants analyzed = participants with available data for VLDL Particles' Size (Small).
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 140
percent change
  week 52 (n = 91) | 49.51 [-41.1 to 140.4]
  week 104 (n = 47) | 30.48 [-75.1 to 136.1]
  week 156 (n = 20) | 9.34 [-48.3 to 67]
  week 208 (n = 19) | -30.36 [-49.8 to -10.9]
  End of treatment (n= 139) | 31.27 [-27.3 to 89.8]
  24 weeks post last dose (n=115) | 32.14 [-5.3 to 69.6]

19. Secondary Outcome: Percent Change From Baseline in Total VLDL Particles' Size and Chylomicron Particles' Size
Description: as for outcome 1
Time Frame: Baseline up to End of treatment; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time. Number of participants analyzed = participants with available data for Total VLDL Particles' Size and Chylomicron Particles' Size.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 140
percent change
  week 52 (n = 91) | 19.94 [-36.7 to 74.6]
  week 104 (n = 47) | -14.25 [-36.4 to 7.9]
  week 156 (n = 20) | 3.48 [-27.5 to 34.5]
  week 208 (n = 19) | -18.66 [-43.6 to 6.3]
  End of treatment (n= 139) | 12.82 [-25.5 to 51.2]
  24 weeks post last dose (n=115) | 19.69 [3.2 to 36.1]

20. Secondary Outcome: Change From Baseline in C-Reactive Protein
Description: as for outcome 1
Time Frame: Baseline up to End of treatment; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 141
percent change
  week 26 (n=130) | 0.67 [-0.8 to 2.1]
  week 52 (n=111) | -0.37 [-1.4 to 0.6]
  week 76 (n=84) | -1.05 [-2 to -0.1]
  week 104 (n=58) | 0.12 [-0.8 to 1]
  week 130 (n=42) | -0.18 [-1.1 to 0.8]
  week 156 (n=30) | 0.02 [-0.5 to 2.1]
  week 182 (n=31) | 0.73 [0.1 to 1.4]
  week 208 (n=27) | 0.2 [-0.5 to 0.9]
  week 234 (n=18) | 0.53 [-0.5 to 1.5]
  End of treatment (n=140) | 0.41 [-0.6 to 1.4]
  24 weeks post last dose (n=116) | 0.09 [-0.9 to 1.1]

21. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1
Description: as for outcome 1
Time Frame: Baseline up to Week 234; 24 weeks post treatment (up to 4.5 years)
Population: Analysis was performed on Safety set. Here n=participants with lipid parameter assessment at specified time.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Mipomersen
Number analyzed (Participants) | 141
percent change
  week 26 (n=130) | -1.01 [-3.8 to 1.7]
  week 52 (n=111) | -1.59 [-4.7 to 1.6]
  week 76 (n=66) | -3.73 [-7.9 to 0.5]
  week 104 (n=57) | -4.33 [-9.1 to 0.4]
  week 130 (n=43) | -1.37 [-6.1 to 3.4]
  week 156 (n=30) | -5.55 [-11.2 to 0]
  week 182 (n=26) | -3.17 [-9.4 to 3.1]
  week 208 (n=27) | -2.19 [-7.2 to 2.8]
  week 234 (n=17) | 3.68 [-3 to 10.3]
  24 weeks post last dose (n = 117) | -0.67 [-3.5 to 2.2]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (59.7 months) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (from the start of study drug in this study up to 24 weeks post-treatment).
Arm/Group | Mipomersen
Serious Adverse Events (participants affected / at risk) | 36/141
Other Adverse Events (participants affected / at risk) | 141/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mipomersen (N=141)
Splenic haemorrhage (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 3
Angina unstable (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 3
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 3
Myocardial infarction (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Device malfunction (General disorders) | 1
Non-cardiac chest pain (General disorders) | 4
Pyrexia (General disorders) | 1
Biliary colic (Hepatobiliary disorders) | 1
Contrast media allergy (Immune system disorders) | 1
Appendicitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amnesia (Nervous system disorders) | 1
Arachnoid cyst (Nervous system disorders) | 1
Dementia Alzheimer's type (Nervous system disorders) | 1
Partial seizures (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Alcoholism (Psychiatric disorders) | 1
Glomerulonephritis membranous (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Ileostomy (Surgical and medical procedures) | 1
Aortic aneurysm (Vascular disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Femoral artery occlusion (Vascular disorders) | 1
Peripheral artery dissection (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mipomersen (N=141)
Anaemia (Blood and lymphatic system disorders) | 9
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Angina pectoris (Cardiac disorders) | 14
Aortic valve disease (Cardiac disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 4
Atrioventricular block second degree (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 2
Extrasystoles (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 4
Supraventricular extrasystoles (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 3
Ventricular dysfunction (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 2
Ear discomfort (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Vertigo (Ear and labyrinth disorders) | 3
Hypothyroidism (Endocrine disorders) | 1
Arcus lipoides (Eye disorders) | 2
Cataract (Eye disorders) | 4
Diplopia (Eye disorders) | 1
Dry eye (Eye disorders) | 2
Eye irritation (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Eyelid cyst (Eye disorders) | 1
Halo vision (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Presbyopia (Eye disorders) | 1
Vision blurred (Eye disorders) | 3
Vitreous floaters (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 14
Abdominal pain lower (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 7
Anal haemorrhage (Gastrointestinal disorders) | 1
Bezoar (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Dental caries (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 21
Diverticulum (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 2
Faecal incontinence (Gastrointestinal disorders) | 1
Faeces soft (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 3
Gastric ulcer (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 4
Gastritis erosive (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Gingival recession (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 2
Hiatus hernia (Gastrointestinal disorders) | 3
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Lip blister (Gastrointestinal disorders) | 1
Lip swelling (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 37
Odynophagia (Gastrointestinal disorders) | 1
Oesophageal dilatation (Gastrointestinal disorders) | 1
Oesophageal spasm (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatic duct dilatation (Gastrointestinal disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Proctitis ulcerative (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Tooth impacted (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 5
Umbilical hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 13
Vomiting projectile (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 6
Chest discomfort (General disorders) | 2
Chest pain (General disorders) | 9
Chills (General disorders) | 27
Cyst (General disorders) | 2
Device breakage (General disorders) | 1
Device failure (General disorders) | 1
Discomfort (General disorders) | 1
Exercise tolerance decreased (General disorders) | 1
Facial pain (General disorders) | 1
Fatigue (General disorders) | 38
Feeling cold (General disorders) | 3
Gait disturbance (General disorders) | 2
Influenza like illness (General disorders) | 70
Injection site atrophy (General disorders) | 1
Injection site bruising (General disorders) | 72
Injection site discolouration (General disorders) | 55
Injection site discomfort (General disorders) | 14
Injection site eczema (General disorders) | 1
Injection site erythema (General disorders) | 117
Injection site exfoliation (General disorders) | 1
Injection site extravasation (General disorders) | 1
Injection site haematoma (General disorders) | 2
Injection site haemorrhage (General disorders) | 17
Injection site hypersensitivity (General disorders) | 2
Injection site hypertrophy (General disorders) | 3
Injection site hypoaesthesia (General disorders) | 2
Injection site induration (General disorders) | 31
Injection site inflammation (General disorders) | 12
Injection site lymphadenopathy (General disorders) | 1
Injection site macule (General disorders) | 4
Injection site mass (General disorders) | 14
Injection site nodule (General disorders) | 9
Injection site oedema (General disorders) | 19
Injection site pain (General disorders) | 102
Injection site pallor (General disorders) | 3
Injection site papule (General disorders) | 7
Injection site paraesthesia (General disorders) | 3
Injection site pruritus (General disorders) | 46
Injection site rash (General disorders) | 16
Injection site reaction (General disorders) | 12
Injection site recall reaction (General disorders) | 10
Injection site swelling (General disorders) | 31
Injection site urticaria (General disorders) | 10
Injection site vesicles (General disorders) | 3
Injection site warmth (General disorders) | 19
Local swelling (General disorders) | 2
Localised oedema (General disorders) | 2
Malaise (General disorders) | 3
Non-cardiac chest pain (General disorders) | 5
Oedema peripheral (General disorders) | 10
Pain (General disorders) | 13
Pyrexia (General disorders) | 25
Swelling (General disorders) | 1
Temperature intolerance (General disorders) | 1
Tenderness (General disorders) | 1
Vaccination site pain (General disorders) | 1
Vessel puncture site bruise (General disorders) | 1
Xerosis (General disorders) | 2
Biliary cyst (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic cyst (Hepatobiliary disorders) | 1
Hepatic fibrosis (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 17
Hepatomegaly (Hepatobiliary disorders) | 9
Hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 3
Serum sickness (Immune system disorders) | 1
Abscess limb (Infections and infestations) | 1
Acarodermatitis (Infections and infestations) | 1
Acute sinusitis (Infections and infestations) | 2
Anal abscess (Infections and infestations) | 1
Asymptomatic bacteriuria (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 10
Bronchopneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Conjunctivitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 4
Eye infection (Infections and infestations) | 2
Folliculitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 4
Gastroenteritis viral (Infections and infestations) | 5
Gastrointestinal infection (Infections and infestations) | 1
Gastrointestinal viral infection (Infections and infestations) | 5
Genital herpes simplex (Infections and infestations) | 1
Giardiasis (Infections and infestations) | 1
H1N1 influenza (Infections and infestations) | 1
Helicobacter gastritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 4
Influenza (Infections and infestations) | 17
Kidney infection (Infections and infestations) | 2
Laryngitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 28
Onychomycosis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 2
Otitis media acute (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 4
Pharyngitis streptococcal (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Post procedural infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 4
Sinobronchitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 20
Skin bacterial infection (Infections and infestations) | 1
Tinea cruris (Infections and infestations) | 1
Tinea versicolour (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 27
Urinary tract infection (Infections and infestations) | 23
Vaginal infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 2
Viral upper respiratory tract infection (Infections and infestations) | 2
Wound infection (Infections and infestations) | 1
Wound sepsis (Infections and infestations) | 2
Animal scratch (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 4
Arthropod sting (Injury, poisoning and procedural complications) | 1
Back injury (Injury, poisoning and procedural complications) | 1
Brain contusion (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 9
Epicondylitis (Injury, poisoning and procedural complications) | 3
Excoriation (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Fractured coccyx (Injury, poisoning and procedural complications) | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 3
Jaw fracture (Injury, poisoning and procedural complications) | 1
Kidney contusion (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 7
Ligament sprain (Injury, poisoning and procedural complications) | 8
Limb injury (Injury, poisoning and procedural complications) | 2
Meniscus injury (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 3
Post procedural contusion (Injury, poisoning and procedural complications) | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 3
Procedural pain (Injury, poisoning and procedural complications) | 9
Procedural vomiting (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Repetitive strain injury (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2
Scratch (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Splenic haematoma (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Suture related complication (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 5
Tibia fracture (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 3
Vaccination complication (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 26
Albumin urine present (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 21
Beta 2 microglobulin urine increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood bicarbonate decreased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 5
Blood phosphorus decreased (Investigations) | 1
Blood potassium increased (Investigations) | 2
Blood pressure increased (Investigations) | 1
Blood testosterone decreased (Investigations) | 1
Blood uric acid increased (Investigations) | 2
Body temperature increased (Investigations) | 2
C-reactive protein increased (Investigations) | 1
Cardiac murmur (Investigations) | 3
Carotid bruit (Investigations) | 4
Electrocardiogram ST segment depression (Investigations) | 1
Electrocardiogram T wave abnormal (Investigations) | 1
Electrocardiogram T wave inversion (Investigations) | 2
Electrocardiogram abnormal (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Haematocrit decreased (Investigations) | 2
Haemoglobin decreased (Investigations) | 2
Heart rate increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 6
International normalised ratio increased (Investigations) | 2
Liver function test abnormal (Investigations) | 3
Liver scan abnormal (Investigations) | 1
Lymph node palpable (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Multiple gated acquisition scan abnormal (Investigations) | 1
Mycobacterium tuberculosis complex test positive (Investigations) | 1
Nuclear magnetic resonance imaging abnormal (Investigations) | 1
Peripheral pulse decreased (Investigations) | 1
Platelet count decreased (Investigations) | 5
Protein urine present (Investigations) | 1
Prothrombin time prolonged (Investigations) | 1
Red blood cell acanthocytes present (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
Red blood cell schistocytes present (Investigations) | 1
Red blood cells urine positive (Investigations) | 2
Scan myocardial perfusion abnormal (Investigations) | 2
Transaminases increased (Investigations) | 1
Urine analysis abnormal (Investigations) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Fluid retention (Metabolism and nutrition disorders) | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 2
Gout (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 19
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 24
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bunion (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 2
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Fracture pain (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 33
Neck pain (Musculoskeletal and connective tissue disorders) | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3
Soft tissue atrophy (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 5
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Burning sensation (Nervous system disorders) | 2
Carotid artery stenosis (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 2
Cluster headache (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 10
Dizziness postural (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 35
Hypoaesthesia (Nervous system disorders) | 7
Lethargy (Nervous system disorders) | 2
Loss of consciousness (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 2
Migraine with aura (Nervous system disorders) | 1
Morton's neuralgia (Nervous system disorders) | 1
Nerve compression (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Orthostatic intolerance (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 4
Post herpetic neuralgia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 2
Restless legs syndrome (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 3
Sinus headache (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 4
Transient ischaemic attack (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 8
VIIth nerve paralysis (Nervous system disorders) | 1
Abnormal sleep-related event (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 6
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 9
Libido decreased (Psychiatric disorders) | 2
Panic attack (Psychiatric disorders) | 1
Stress (Psychiatric disorders) | 2
Albuminuria (Renal and urinary disorders) | 1
Bladder discomfort (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 4
Haematuria (Renal and urinary disorders) | 6
Micturition urgency (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Nephropathy (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 4
Proteinuria (Renal and urinary disorders) | 6
Pyelocaliectasis (Renal and urinary disorders) | 1
Pyuria (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 4
Renal failure (Renal and urinary disorders) | 1
Stress urinary incontinence (Renal and urinary disorders) | 1
Urge incontinence (Renal and urinary disorders) | 1
Urinary tract disorder (Renal and urinary disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1
Breast mass (Reproductive system and breast disorders) | 2
Dyspareunia (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Menopausal symptoms (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Menstruation delayed (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Pruritus genital (Reproductive system and breast disorders) | 1
Testicular cyst (Reproductive system and breast disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Blister (Skin and subcutaneous tissue disorders) | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 3
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 3
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Ingrown hair (Skin and subcutaneous tissue disorders) | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 1
Macule (Skin and subcutaneous tissue disorders) | 2
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 6
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 1
Scab (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2
Skin plaque (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 6
Xanthelasma (Skin and subcutaneous tissue disorders) | 2
Xanthoma (Skin and subcutaneous tissue disorders) | 1
Aortic aneurysm (Vascular disorders) | 3
Aortic arteriosclerosis (Vascular disorders) | 1
Aortic calcification (Vascular disorders) | 1
Aortic dilatation (Vascular disorders) | 3
Aortic stenosis (Vascular disorders) | 1
Flushing (Vascular disorders) | 3
Haematoma (Vascular disorders) | 2
Hot flush (Vascular disorders) | 4
Hypertension (Vascular disorders) | 8
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Infarction (Vascular disorders) | 1
Intermittent claudication (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Pallor (Vascular disorders) | 1
Peripheral coldness (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Subclavian artery stenosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.